CLINICAL TRIAL: NCT00597831
Title: Regulation of Intracerebral Pressure During Electroconvulsive Therapy. Does Systemic Bloodpressure Reflect the Intracranial Pressure?
Brief Title: Regulation of Intracerebral Pressure During Electroconvulsive Therapy
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Derikx, MD, Rijnstate Hospital
Other Study IDs: LTC-491/251007
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Depression; Intracranial Pressure
Keywords: depression; electroconvulsive therapy; Ultrasonography Doppler Transcranial; intracranial pressure
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: All patients in the Rijnstate Hospital with an indication for unilateral ECT treatment and a major depression or psychotic depression according to DSM IV-TR criteria.

SUMMARY:
The purpose of this study is to determine whether electroconvulsive therapy (ECT) has an influence on pressure within the human brain before, during and after ECT.

DETAILED DESCRIPTION:
1. Aim:

   1. Our main objective concerning this study is to determine to what extent ECT does lead to an increase of the Pulsatility Index (as an indicator of intracerebral pressure) measured by a Transcranial Doppler Device (TCD).
   2. As a secondary objective we want to compare the PI measurements with simultaneously measured systemic blood pressure.
2. Study design:

   a.Observational study: cohort study
3. Treatment:

   a. Treatment as usual, PI and blood pressure measurement at baseline, just before ECT, during and 5 minutes after ECT. Data will be collected during unilateral treatment during 3 consecutive ECT treatments.
4. Endpoints:

   1. A minimum of sixteen patients are needed according to the power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Temporal window to measure PI
* Major depression
* Psychotic depression

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients indicated for unilateral ECT treatment in the Rijnstate Hospital with the diagnosis major depression and psychotic depressionaccording to DSM IV-TR classification. Patients who already started treatment and patients just starting ECT and are of age > 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pulsatility Index before, during and after electroconvulsive therapy | before, during and after three consecutive ECT treatments

SECONDARY OUTCOMES:
Bloodpressure before, during and after ECT. | before, during and after three consecutive ECT treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Roy LE Derikx, MD, Principal Investigator — Rijnstate Hospital
Locations (1):
- PAAZ Rijnstate Hospital, Arnhem, Gelderland, Netherlands